CLINICAL TRIAL: NCT04057573
Title: Topical Ruxolitinib Evaluation in Vitiligo Study 2 (TRuE-V2): A Phase 3, Double-Blind, Randomized, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream Followed by an Extension Period in Participants With Vitiligo
Brief Title: Topical Ruxolitinib Evaluation in Vitiligo Study 2 (TRuE-V2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-307; 2019-000847-28 (EudraCT Number)
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Non-segmental Vitiligo
Keywords: Vitiligo; non-segmental; JAK inhibitor
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: Participants will receive ruxolitinib cream or vehicle for 24 weeks, after which they will be offered the opportunity to continue in the treatment extension period. Participants initially randomized to vehicle will be crossed over to active drug, and participants treated with ruxolitinib cream will receive an additional 28 weeks of treatment with ruxolitinib cream.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind Period: Ruxolitinib cream 1.5% BID (Experimental): Participants applied ruxolitinib 1.5% cream twice daily (BID) for 24 weeks.
  Interventions: Drug: Ruxolitinib cream
- Double-Blind Period: Vehicle cream BID (Placebo Comparator): Participants applied matching vehicle cream BID for 24 weeks.
  Interventions: Drug: Vehicle
- Treatment-Extension Period: Ruxolitinib cream 1.5% BID (Experimental): Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-Blind Period continued to apply ruxolitinib cream 1.5% BID for an additional 28 weeks in the Treatment-Extension Period.
  Interventions: Drug: Ruxolitinib cream
- Treatment-Extension Period: Vehicle cream to Ruxolitinib cream 1.5% BID (Experimental): Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied vehicle cream BID during the Double-Blind Period applied ruxolitinib cream 1.5%m BID for 28 weeks in the Treatment-Extension Period.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB018424 cream
  Arms: Double-Blind Period: Ruxolitinib cream 1.5% BID; Treatment-Extension Period: Ruxolitinib cream 1.5% BID; Treatment-Extension Period: Vehicle cream to Ruxolitinib cream 1.5% BID
Drug: Vehicle — Vehicle cream is a topical formulation applied as a thin film to affected areas.
  Arms: Double-Blind Period: Vehicle cream BID; Treatment-Extension Period: Vehicle cream to Ruxolitinib cream 1.5% BID

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in adolescent and adult participants with non-segmental vitiligo for whom total body involved vitiligo area (facial and nonfacial) does not exceed 10% body surface area (BSA).

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of non-segmental vitiligo with depigmented area including ≥ 0.5% BSA on the face, ≥ 0.5 F-VASI, ≥ 3% BSA on nonfacial areas, ≥ 3 T-VASI, and total body vitiligo area (facial and nonfacial) not exceeding 10% BSA.
* Agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit. Over-the-counter preparations deemed acceptable by the investigator and camouflage makeups are permitted.
* Must be willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child for the duration of study participation.

Key Exclusion Criteria:

* No pigmented hair within any of the vitiligo areas on the face.
* Other forms of vitiligo (eg, segmental) or other differential diagnosis of vitiligo or other skin depigmentation disorders (eg, piebaldism, pityriasis alba, leprosy, postinflammatory hypopigmentation, progressive macule hypomelanosis, nevus anemicus, chemical leukoderma, and tinea versicolor).
* Have used depigmentation treatments (eg, monobenzone) for past treatment of vitiligo or other pigmented areas.
* Use of protocol-defined treatments within the indicated washout period before baseline.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (74):
- United States (33):
  - Desert Sky Dermatology, Gilbert, Arizona
  - Center For Dermatology Cosmetic and Laser Surgery, Fremont, California
  - Uci Beckman Laser Institute and Medical Clinic, Irvine, California
  - UCI Health Beckman Laser Institute and Medical Center, Irvine, California
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists Inc, Murrieta, California
  - Dermatology Specialists Inc, Oceanside, California
  - Integrative Skin Science and Research, Sacramento, California
  - Acrc Studies, San Diego, California
  - Central Sooner Research, San Diego, California
  - Colorado Medical Research Center Inc, Denver, Colorado
  - Advanced Pharma Cr, Miami, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - Avita Clinical Research, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Ashira Dermatology Llc, Gurnee, Illinois
  - Randall Dermatology of West Lafayette, West Lafayette, Indiana
  - Randall Dermatology, West Lafayette, Indiana
  - Delricht Clinical Research - Clinedge - Ppds Baton Rouge, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Minnesota Clinical Study Center, Minneapolis, Minnesota
  - Jdr Dermatology Research, Las Vegas, Nevada
  - Northwell Physician Partners, New Hyde Park, New York
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Derm Research Center of New York Inc, Stony Brook, New York
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Clinical Research Partners Llc, Richmond, Virginia
- Bulgaria (7):
  - Medical Center Unimed Eood, Sevlievo
  - Medical Center Unimed EOOD, Sevlievo
  - Diagnostic Consultative Center Ii Sofia Eood, Sofia
  - University Multiprofile Hospital For Active Treatment Aleksandrovska, Sofia
  - Diagnostic Consultative Center II Sofia EOOD, Sofia
  - University Hospital Prof Dr Stoyan Kirkovich, Stara Zagora
  - University Hospital " Prof. Dr Stoyan Kirkovich", Stara Zagora
- Canada (5):
  - Simcoderm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Xlr8 Medical Research, Windsor, Ontario
- France (7):
  - Centre Hospitalier Universitaire de Besancon, Besançon
  - CHU Besancon, Besançon
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - CHU de Bordeaux, Hospital Saint Andre, Bordeaux
  - University Hospital Henri Mondor, Créteil
  - CENTRE HOSpITALIER UNIVERSITAIRE HENRI MONDOR, Créteil
  - Le Bateau Blanc, Martigues
- Germany (5):
  - Emovis GMBH, Berlin
  - Universitatsklinikum Bonn Aoer, Bonn
  - Hautarztpraxis Mahlow, Mahlow
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - University Medical Center (Universitätsmedizin der Johannes Gutenberg-Universität Mainz), Mainz
- Italy (2):
  - Policlinico S. Orsola Malpighi, Bologna
  - Istituto Dermatologico San Gallicano, Rome
- Amsterdam University Medical Centre, Amsterdam, Netherlands
- Poland (8):
  - Synexus Polska Sp. Z o.o. Oddział w Częstochowie, Częstochowa
  - Synexus Affiliate - Krakowskie Centrum Medyczne, Krakow
  - Synexus Polska Sp Z Oo Oddzial W Lodzi, Lodz
  - Synexus Polska Sp Z Oo Oddzial W Czestochowie, Lublin
  - Lubeskie Centrum Diagnostyczne, Świdnik
  - Synexus Polska Sp. Z O.O. Oddzial Warszawie, Warsaw
  - High-Med Przychodnia Specjalistycza, Warsaw
  - Dermmedica Sp. Z O.O., Wroclaw
- Spain (6):
  - Ico Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Dermomedic, Madrid
  - IDEI (Instituto de Dermatología Integral)., Madrid
  - Hospital La Paz (Hospital Universitario La Paz ), Madrid
  - Hospital Universitario de La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosmarin D, Pandya AG, Passeron T, Forman SB, Zdybski J, Amster M, Feser C, Papp KA, Nuara A, Kornacki D, Wei S, Ren H, Harris JE, Ezzedine K. Long-Term Integrated Safety Summary of Ruxolitinib Cream in Phase 3 Clinical Trials of Patients with Vitiligo. Dermatol Ther (Heidelb). 2025 Dec;15(12):3703-3716. doi: 10.1007/s13555-025-01555-3. Epub 2025 Oct 22. PMID 41125994
- [Derived] Seneschal J, Wolkerstorfer A, Desai SR, Grimes P, Ezzedine K, Pandya AG, Kornacki D, Wei S, Passeron T, Rosmarin D. Efficacy and Safety of Ruxolitinib Cream in Vitiligo by Patient Characteristic Subgroups: Descriptive Pooled Analysis From Two Phase 3 Studies. Dermatol Ther (Heidelb). 2025 May;15(5):1227-1238. doi: 10.1007/s13555-025-01381-7. Epub 2025 Mar 29. PMID 40156697
- [Derived] Bibeau K, Butler K, Wang M, Skaltsa K, Hamzavi IH. Psychometric Evaluation of the Facial and Total Vitiligo Area Scoring Index Instruments in the TRuE-V Phase 3 Studies. Dermatol Ther (Heidelb). 2024 Aug;14(8):2223-2234. doi: 10.1007/s13555-024-01223-y. Epub 2024 Jul 30. PMID 39078582
- [Derived] Rosmarin D, Passeron T, Pandya AG, Grimes P, Harris JE, Desai SR, Lebwohl M, Ruer-Mulard M, Seneschal J, Wolkerstorfer A, Kornacki D, Sun K, Butler K, Ezzedine K; TRuE-V Study Group. Two Phase 3, Randomized, Controlled Trials of Ruxolitinib Cream for Vitiligo. N Engl J Med. 2022 Oct 20;387(16):1445-1455. doi: 10.1056/NEJMoa2118828. PMID 36260792
- See also: Plain Language Summary for Upload to Incyteclinicaltrials.com — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217471&parentIdentifier=INCB%2018424-307&attachmentIdentifier=236ef937-0530-4f1d-98dd-3b1a5e0f683c&fileName=Incyte_PLS_INCB18424-307_Final.19_December_2023.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 49 study centers in North America and Europe.
Pre-assignment Details: A total of 344 participants were randomized into the study. Of the 344 randomized participants (Intent-to-Treat Population), 343 applied study drug at least once (Safety Population); 297 participants applied ruxolitinib cream at least once during the Treatment-Extension (TE) Period (TE Evaluable Population).
Period: 24-Week Double-Blind Period
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 229 | 115 | 0 | 0
ITT Population | 229 | 115 | 0 | 0
ITT Population, Excluding Non-compliant Site | 222 | 109 | 0 | 0
Completed | 199 | 98 | 0 | 0
Not Completed | 30 | 17 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 11 | 6 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 8 | 0 | 0
Not completed — Discontinued Treatment due to COVID-19 Pandemic | 3 | 1 | 0 | 0
Not completed — Non-compliance with Attending Study Visits | 1 | 0 | 0 | 0
Not completed — Unable to Attend Study Visits Due to Travel | 0 | 1 | 0 | 0
Not completed — Not Treated | 1 | 0 | 0 | 0
Period: 28-Week Treatment Extension Period
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 0 | 0 | 199 (Treatment-Extension Evaluable Population: all participants who applied ruxolitinib cream at least once in the TE period) | 98
Completed | 0 | 0 | 178 | 79
Not Completed | 0 | 0 | 21 | 19
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 9 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 9
Not completed — Unable to Perform Safety Follow-up Visit | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all participants who applied ruxolitinib cream or vehicle cream at least once. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Total
Number analyzed (Participants) | 228 | 115 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (15.22) | 39.8 (12.12) | 38.9 (14.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 60 | 172
  Male | 116 | 55 | 171
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 182 | 93 | 275
  Black/African American | 12 | 5 | 17
  Asian | 12 | 7 | 19
  American Indian/Alaska Native | 1 | 0 | 1
  Native Hawaiian/Pacific Islander | 2 | 0 | 2
  Not Reported | 3 | 3 | 6
  North African | 2 | 0 | 2
  White/Caucasian and Asian | 1 | 0 | 1
  Guyana | 1 | 0 | 1
  Cape Verdean | 1 | 1 | 2
  Persian | 1 | 0 | 1
  Middle Eastern | 3 | 0 | 3
  Arab/North-African | 1 | 0 | 1
  White/Black/Asian | 1 | 0 | 1
  Mexican | 2 | 1 | 3
  Jordanian | 1 | 0 | 1
  Arabic | 1 | 0 | 1
  Argentinian | 1 | 0 | 1
  Brazilian | 0 | 2 | 2
  Dominican Republic | 0 | 1 | 1
  Indo-Caribbean | 0 | 1 | 1
  Multi-National | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 32 | 82
  Not Hispanic or Latino | 174 | 80 | 254
  Not Reported | 2 | 3 | 5
  Captured as "Other" | 2 | 0 | 2
Face Vitiligo Area Scoring Index (F-VASI) [Mean (Standard Deviation); unit: scores on a scale] — F-VASI was measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]; assessed by the Investigator) and the degree of depigmentation: 0% (no depigmentation), 10% (specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), 100% (no pigment). F-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each facial site and summing all values (range: 0-3; higher values=worse outcome).
  scores on a scale | 0.900 (0.5248) | 0.834 (0.5233) | 0.878 (0.5245)
Facial Body Surface Area (F-BSA) Involvement [Mean (Standard Deviation); unit: percentage of facial surface area] — F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids.
  percentage of facial surface area | 0.98 (0.570) | 0.92 (0.569) | 0.96 (0.569)
Total Body Vitiligo Area Scoring Index (T-VASI) [Mean (Standard Deviation); unit: scores on a scale] — T-VASI was measured by the percentage of vitiligo involvement from all body regions (percentage of BSA; Investigator assessed) and the degree of depigmentation: 0% (no depigmentation), 10% (specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), 100% (no pigment). T-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each site and summing all values (possible range: 0-100; higher values=worse outcome).
  scores on a scale | 6.844 (2.0574) | 7.022 (2.1986) | 6.904 (2.1043)
Total Body Surface Area (T-BSA) Involvement [Mean (Standard Deviation); unit: percentage of total body surface area] — T-BSA involvement was the proportion of the body surface area with vitiligo. The body was divided into the following 6 separate and mutually exclusive sites: (1) head/neck, (2) hands, (3) upper extremities (excluding hands), (4) trunk, (5) lower extremities (excluding feet), and (6) feet.
  percentage of total body surface area | 7.44 (2.011) | 7.68 (2.040) | 7.52 (2.021)
Age Continuous, without Noncompliant Site [Mean (Standard Deviation); unit: years] — Population: Baseline data are reported for members of the Intent-to-Treat (ITT) Population (all randomized participants), minus those participants enrolled at the noncompliant site. Treatment groups for this population were defined according to the treatment assignment at the time of randomization).
  years
    number analyzed (Participants) | 222 | 109 | 331
    (all) | 38.4 (15.44) | 39.4 (12.29) | 38.7 (14.46)
Gender, without Noncompliant Site [Count of Participants; unit: Participants] — Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  Participants
    Female: number analyzed (Participants) | 222 | 109 | 331
    Female | 110 | 58 | 168
    Male: number analyzed (Participants) | 222 | 109 | 331
    Male | 112 | 51 | 163
Race, without Noncompliant Site [Count of Participants; unit: Participants] — Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  Participants
    White: number analyzed (Participants) | 222 | 109 | 331
    White | 178 | 88 | 266
    Black/African American: number analyzed (Participants) | 222 | 109 | 331
    Black/African American | 11 | 5 | 16
    Asian: number analyzed (Participants) | 222 | 109 | 331
    Asian | 11 | 6 | 17
    American Indian/Alaska Native: number analyzed (Participants) | 222 | 109 | 331
    American Indian/Alaska Native | 1 | 0 | 1
    Native Hawaiian/Pacific Islander: number analyzed (Participants) | 222 | 109 | 331
    Native Hawaiian/Pacific Islander | 2 | 0 | 2
    Not Reported: number analyzed (Participants) | 222 | 109 | 331
    Not Reported | 3 | 3 | 6
    North African: number analyzed (Participants) | 222 | 109 | 331
    North African | 2 | 0 | 2
    White/Caucasian and Asian: number analyzed (Participants) | 222 | 109 | 331
    White/Caucasian and Asian | 1 | 0 | 1
    Guyana: number analyzed (Participants) | 222 | 109 | 331
    Guyana | 1 | 0 | 1
    Cape Verdean: number analyzed (Participants) | 222 | 109 | 331
    Cape Verdean | 1 | 1 | 2
    Persian: number analyzed (Participants) | 222 | 109 | 331
    Persian | 1 | 0 | 1
    Middle Eastern: number analyzed (Participants) | 222 | 109 | 331
    Middle Eastern | 3 | 0 | 3
    Arab/North-African: number analyzed (Participants) | 222 | 109 | 331
    Arab/North-African | 1 | 0 | 1
    White/Black/Asian: number analyzed (Participants) | 222 | 109 | 331
    White/Black/Asian | 1 | 0 | 1
    Mexican: number analyzed (Participants) | 222 | 109 | 331
    Mexican | 2 | 1 | 3
    Jordanian: number analyzed (Participants) | 222 | 109 | 331
    Jordanian | 1 | 0 | 1
    Arabic: number analyzed (Participants) | 222 | 109 | 331
    Arabic | 1 | 0 | 1
    Argentinian: number analyzed (Participants) | 222 | 109 | 331
    Argentinian | 1 | 0 | 1
    Brazilian: number analyzed (Participants) | 222 | 109 | 331
    Brazilian | 0 | 2 | 2
    Dominican Republic: number analyzed (Participants) | 222 | 109 | 331
    Dominican Republic | 0 | 1 | 1
    Indo-Caribbean: number analyzed (Participants) | 222 | 109 | 331
    Indo-Caribbean | 0 | 1 | 1
    Multi-National: number analyzed (Participants) | 222 | 109 | 331
    Multi-National | 0 | 1 | 1
Ethnicity, without Noncompliant Site [Count of Participants; unit: Participants] — Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 222 | 109 | 331
    Hispanic or Latino | 49 | 30 | 79
    Not Hispanic or Latino: number analyzed (Participants) | 222 | 109 | 331
    Not Hispanic or Latino | 169 | 76 | 245
    Not Reported: number analyzed (Participants) | 222 | 109 | 331
    Not Reported | 2 | 3 | 5
    Captured as "Other": number analyzed (Participants) | 222 | 109 | 331
    Captured as "Other" | 2 | 0 | 2
F-VASI, without Noncompliant Site [Mean (Standard Deviation); unit: scores on a scale] — F-VASI was measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]; assessed by the Investigator) and the degree of depigmentation: 0% (no depigmentation), 10% (specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), 100% (no pigment). F-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each facial site and summing all values (range: 0-3; higher values=worse outcome). Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  scores on a scale
    number analyzed (Participants) | 222 | 109 | 331
    (all) | 0.898 (0.5256) | 0.834 (0.5342) | 0.877 (0.5285)
F-BSA Involvement, without Noncompliant Site [Mean (Standard Deviation); unit: percentage of facial surface area] — F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  percentage of facial surface area
    number analyzed (Participants) | 222 | 109 | 331
    (all) | 0.98 (0.571) | 0.92 (0.582) | 0.96 (0.575)
T-VASI, without Noncompliant Site [Mean (Standard Deviation); unit: scores on a scale] — T-VASI was measured by the percentage of vitiligo involvement from all body regions (percentage of BSA; Investigator assessed) and the degree of depigmentation: 0% (no depigmentation), 10% (specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), 100% (no pigment). T-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each site and summing all values (possible range: 0-100; higher values=worse outcome). Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  scores on a scale
    number analyzed (Participants) | 222 | 109 | 331
    (all) | 6.790 (2.0435) | 6.979 (2.1953) | 6.852 (2.0933)
T-BSA Involvement, without Noncompliant Site [Mean (Standard Deviation); unit: percentage of total body surface area] — T-BSA involvement was the proportion of the body surface area with vitiligo. The body was divided into the following 6 separate and mutually exclusive sites: (1) head/neck, (2) hands, (3) upper extremities (excluding hands), (4) trunk, (5) lower extremities (excluding feet), and (6) feet. Population: Baseline data are reported for members of the ITT Population, minus those participants enrolled at the noncompliant site.
  percentage of total body surface area
    number analyzed (Participants) | 222 | 109 | 331
    (all) | 7.38 (2.025) | 7.66 (2.040) | 7.47 (2.031)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a ≥ 75% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI75) Score at Week 24
Description: An F-VASI75 responder achieved at least 75% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: Intent-to-Treat Population: all randomized participants. Treatment groups for this population were defined according to the treatment assignment at the time of randomization. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Missing F-VASI scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors as predicators.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants | 30.9 | 11.4
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p = 0.0004, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 3.45, 95% CI 2-sided [1.737 to 6.835]

2. Secondary Outcome: Percentage of Participants Achieving a ≥ 50% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI50) Score at Week 24
Description: An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Missing F-VASI scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors as predicators.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants | 51.4 | 20.9
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p < 0.0001, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 3.99, 95% CI 2-sided [2.296 to 6.949]

3. Secondary Outcome: Percentage of Participants Achieving a ≥ 90% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI90) Score at Week 24
Description: An F-VASI90 responder achieved at least 90% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants | 16.3 | 1.3
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p = 0.0065, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 15.29, 95% CI 2-sided [2.150 to 108.739]

4. Secondary Outcome: Percentage of Participants Achieving a ≥ 50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) Score at Week 24
Description: A T-VASI50 responder achieved at least 50% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to the nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Missing T-VASI scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors as predicators.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants | 23.9 | 6.8
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p = 0.0006, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 4.29, 95% CI 2-sided [1.865 to 9.853]

5. Secondary Outcome: Percentage of Participants Achieving a Vitiligo Noticeability Scale (VNS) of 4 or 5 at Week 24
Description: The VNS is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. The Baseline facial photograph was shown to the participants for reference, and a mirror was provided for the participants to assess the vitiligo on their face. The participant was asked to respond to the following query: Compared with before treatment, how noticeable is the vitiligo now? Responses: (1) more noticeable, (2) as noticeable, (3) slightly less noticeable, (4) a lot less noticeable, and (5) no longer noticeable.
Time Frame: Baseline; Week 24
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Missing VNS scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors as predicators.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants | 20.5 | 4.9
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p = 0.0013, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 4.86, 95% CI 2-sided [1.851 to 12.755]

6. Secondary Outcome: Percentage Change From Baseline in Facial Body Surface Area (F-BSA) at Week 24
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline (BL) value minus BL value]/BL value) X 100.
Time Frame: Baseline; Week 24
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Missing F-BSA scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors as predicators.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage change | -26.4 (2.57) | -7.0 (3.82)
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p < 0.0001, ANCOVA — Response Variable = Treatment + Stratification Factors (Skin Type Fitzpatrick scale Type I, II versus Type III, IV, V, and VI, Region North America/Europe) + Baseline; Least squares mean difference = -19.5, 95% CI 2-sided [-28.46 to -10.45], Standard Error of Mean 4.59

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Double-Blind Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 24)
Population: Safety Population: all participants who applied ruxolitinib cream or vehicle cream at least once. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 228 | 115
Participants | 114 | 39

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Treatment-Extension Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from the completion of the Week 24 assessments until at least 30 days after the last application of study drug (up to Week 52 + 30 days)
Population: Treatment-Extension (TE) Evaluable Population: all participants who applied ruxolitinib cream at least once in the TE Period
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 199 | 98
Participants | 82 | 38

9. Secondary Outcome: Percentage of Participants Achieving a ≥ 25% Improvement in the Face Vitiligo Area Scoring Index (F-VASI25) Score at Week 24
Description: An F-VASI25 responder achieved at least 25% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants | 63.9 | 32.0
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p < 0.0001, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 3.76, 95% CI 2-sided [2.267 to 6.246]

10. Secondary Outcome: Percentage of Participants Achieving a ≥ %25, ≥ %50, ≥ 75%, and ≥ 90% Improvement in the Face Vitiligo Area Scoring Index (F-VASI25/50/75/90) Score at Week 52
Description: An F-VASI25/50/75/90 responder achieved at least 25/50/75/90% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Week 52
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 177 | 81
percentage of participants
  F-VASI25 | 82.5 | 71.6
  F-VASI50 | 74.0 | 49.4
  F-VASI75 | 48.0 | 29.6
  F-VASI90 | 27.7 | 16.0

11. Secondary Outcome: Percentage Change From Baseline in F-VASI at Week 24
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; Week 24
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Only participants with available data were analyzed. MMRM model: (Response Variable = Treatment + Stratification Factors [Skin Type Fitzpatrick Scale Type I and II versus Type III, IV, V, and VI, Region North America/Europe] + Visit + Treatment*Visit).
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 199 | 98
percentage change | -44.39 (2.85) | -15.80 (4.04)
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p < 0.0001, mixed-effect model; repeated measurement; Least squares mean difference = -28.59, 95% CI 2-sided [-38.33 to -18.86], Standard Error of Mean 4.94

12. Secondary Outcome: Percentage Change From Baseline in F-VASI at Week 52
Description: as for outcome 11
Time Frame: Baseline; Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 177 | 81
percentage change | -63.75 (34.103) | -43.50 (47.509)

13. Secondary Outcome: Percentage Change From Baseline in F-BSA at Week 52
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 177 | 81
percentage change | -41.81 (35.694) | -23.45 (46.360)

14. Secondary Outcome: Percentage Change From Baseline in T-VASI at Week 24
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to the nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; Week 24
Population: ITT Population. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Only participants with available data were analyzed. MMRM model: (Response Variable = Treatment + Stratification Factors [Skin Type Fitzpatrick scale Type I and II vs Type III, IV, V, and VI, Region North America/Europe] + Visit + Treatment*Visit).
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 199 | 98
percentage change | -28.85 (1.96) | -8.99 (2.78)
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p < 0.0001, mixed-effect model; repeated measurement; least squares mean difference = -19.85, 95% CI 2-sided [-26.55 to -13.16], Standard Error of Mean 3.40

15. Secondary Outcome: Percentage Change From Baseline in T-VASI at Week 52
Description: as for outcome 14
Time Frame: Baseline; Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 177 | 81
percentage change | -46.80 (29.903) | -30.11 (30.315)

16. Secondary Outcome: Percentage Change From Baseline in T-BSA at Week 24
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 199 | 98
percentage change | -14.23 (1.55) | -2.28 (2.19)
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p < 0.0001, mixed-effect model; repeated measurement; least squares mean difference = -11.95, 95% CI 2-sided [-17.23 to -6.67], Standard Error of Mean 2.68

17. Secondary Outcome: Percentage Change From Baseline in T-BSA at Week 52
Description: as for outcome 16
Time Frame: Baseline; Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 177 | 81
percentage change | -26.04 (28.481) | -13.54 (27.144)

18. Secondary Outcome: Percentage of Participants Achieving a ≥ 25%, ≥ 75%, and ≥ 90% Improvement in the Total Body Vitiligo Area Scoring Index (T-VASI25/75/90) Score at Week 24
Description: A T-VASI25/75/90 responder achieved at least 25/75/90% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 222 | 109
percentage of participants
  T-VASI25 | 50.2 | 21.2
  T-VASI75 | 8.0 | 1.8
  T-VASI90 | 1.0 | 0.0
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; T-VASI25; Test type: Superiority; p < 0.0001, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 3.75, 95% CI 2-sided [2.121 to 6.630]
Statistical Analysis 2: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; T-VASI75; Test type: Superiority; p = 0.0436, exact logistic regression — The model included the treatment group (1.5% BID and vehicle) and stratification factors (skin type and region); Odds Ratio (OR) = 4.59, 95% CI 2-sided [1.045 to 20.192]
Statistical Analysis 3: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; T-VASI90; Test type: Superiority; The p value was not evaluable because the response rate in the vehicle group was too low; Odds Ratio (OR) = 1.35

19. Secondary Outcome: Percentage of Participants Achieving a ≥ 25%, ≥ 50%, ≥ 75%, and ≥ 90% Improvement in the Total Body Vitiligo Area Scoring Index (T-VASI25/50/75/90) Score at Week 52
Description: A T-VASI25/50/75/90 responder achieved ≥25/50/75/90% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; Week 52
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 177 | 81
percentage of participants
  T-VASI25 | 76.8 | 53.1
  T-VASI50 | 49.2 | 22.2
  T-VASI75 | 20.9 | 8.6
  T-VASI90 | 6.8 | 1.2

20. Secondary Outcome: Percentage of Participants in Each Category of VNS During the Treatment Period (Double-Blind and Treatment-Extension Periods)
Description: as for outcome 5
Time Frame: Baseline; Week 24 and Week 52
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 199 | 98 | 177 | 81
percentage of participants
  Week 24, more noticeable: number analyzed (Participants) | 199 | 98 | 0 | 0
  Week 24, more noticeable | 8.5 | 11.2 |  |
  Week 24, as noticeable: number analyzed (Participants) | 199 | 98 | 0 | 0
  Week 24, as noticeable | 30.7 | 58.2 |  |
  Week 24, slightly less noticeable: number analyzed (Participants) | 199 | 98 | 0 | 0
  Week 24, slightly less noticeable | 40.2 | 25.5 |  |
  Week 24, a lot less noticeable: number analyzed (Participants) | 199 | 98 | 0 | 0
  Week 24, a lot less noticeable | 20.6 | 4.1 |  |
  Week 24, no longer noticeable: number analyzed (Participants) | 199 | 98 | 0 | 0
  Week 24, no longer noticeable | 0.0 | 1.0 |  |
  Week 52, more noticeable: number analyzed (Participants) | 0 | 0 | 177 | 81
  Week 52, more noticeable |  |  | 4.5 | 11.1
  Week 52, as noticeable: number analyzed (Participants) | 0 | 0 | 177 | 81
  Week 52, as noticeable |  |  | 16.4 | 25.9
  Week 52, slightly less noticeable: number analyzed (Participants) | 0 | 0 | 177 | 81
  Week 52, slightly less noticeable |  |  | 46.3 | 49.4
  Week 52, a lot less noticeable: number analyzed (Participants) | 0 | 0 | 177 | 81
  Week 52, a lot less noticeable |  |  | 32.2 | 13.6
  Week 52, no longer noticeable: number analyzed (Participants) | 0 | 0 | 177 | 81
  Week 52, no longer noticeable |  |  | 0.6 | 0.0

21. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 24
Description: The DLQI is a 10-question validated questionnaire for use in participants aged 16 years and over to measure how much the skin problem has affected the participant over the previous 7 days. Each question is scored as: very much = 3; a lot = 2; a little = 1; not at all = 0; not relevant = 0. For Question 7, "Prevented work or studying" = 3. The DLQI was calculated by summing the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline; Week 24
Population: ITT Population: participants aged ≥ 16 years. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Only participants with available data were analyzed. MMRM model: (Response Variable = Treatment + Stratification Factors [Skin Type Fitzpatrick scale Type I and II vs Type III, IV, V, and VI, Region North America/Europe] + Visit + Treatment*Visit).
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 182 | 94
scores on a scale | -1.19 (0.30) | -0.59 (0.41)
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID vs Double-Blind Period: Vehicle Cream BID; Test type: Superiority; p = 0.2350, mixed-effect model; repeated measurement; least squares mean difference = -0.60, 95% CI 2-sided [-1.60 to 0.39], Standard Error of Mean 0.51

22. Secondary Outcome: Change From Baseline in DLQI at Week 52
Description: as for outcome 21
Time Frame: Baseline; Week 52
Population: ITT Population: participants aged ≥ 16 years. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 205 | 105
scores on a scale
  Baseline | 4.37 (4.485) | 5.38 (4.876)
  Week 52: number analyzed (Participants) | 161 | 78
  Week 52 | -0.84 (3.976) | -1.15 (4.264)

23. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) During the Treatment Period (Double-Blind and Treatment-Extension Periods)
Description: The DLQI is a 10-question validated questionnaire for use in participants aged 16 years and over to measure how much the skin problem has affected the participant over the previous 7 days. The CDLQI is the youth/children's version of the DLQI and was completed by adolescents aged ≥ 12 years to < 16 years. Each question is scored as: very much = 3; quite a lot = 2; only a little = 1; not at all = 0; question unanswered = 0. For Question 7: "Prevented school" = 3. The CDLQI was calculated by summing the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline; Week 24 and Week 52
Population: ITT Population: participants aged < 16 years. Data from participants at a single site were excluded from this analysis owing to serious noncompliance with the protocol. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 17 | 3 | 16 | 3
scores on a scale
  Baseline: number analyzed (Participants) | 17 | 3 | 0 | 0
  Baseline | 1.29 (2.201) | 6.33 (10.116) |  |
  Week 24: number analyzed (Participants) | 17 | 3 | 0 | 0
  Week 24 | 0.00 (1.837) | -2.33 (8.505) |  |
  Week 52: number analyzed (Participants) | 0 | 0 | 16 | 3
  Week 52 |  |  | 1.19 (4.665) | -1.00 (4.583)

24. Secondary Outcome: Trough Plasma Concentrations of Ruxolitinib at Weeks 4, 24, and 40
Description: Trough plasma concentration was defined as the measurement of the plasma concentration of ruxolitinib before drug application.
Time Frame: pre-dose at Weeks 4, 24, and 40
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) Evaluable Population: all participants who applied ruxolitinib cream at least once and provided at least 1 postdose blood sample that complied with the Protocol
Measure: Mean (Standard Deviation); unit: nanomoles
Groups:
- Ruxolitinib Cream: Participants received ruxolitinib cream 1.5% twice daily (BID) for 24 weeks, followed by ruxolitinib cream 1.5% BID for an additional 28-week treatment extension period.
Arm/Group | Ruxolitinib Cream | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 208 | 0 | 184 | 83
nanomoles
  Week 4: number analyzed (Participants) | 208 | 0 | 0 | 0
  Week 4 | 61.0 (68.6) |  |  |
  Week 24: number analyzed (Participants) | 208 | 0 | 0 | 0
  Week 24 | 54.5 (79.1) |  |  |
  Week 40: number analyzed (Participants) | 0 | 0 | 184 | 83
  Week 40 |  |  | 57.0 (73.3) | 48.2 (57.0)

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 52 + 30 days)
Description: Treatment-emergent adverse events (TEAEs): AEs reported for the first time or the worsening of a pre-existing event after the first application of study drug. For the Double-Blind Period, TEAEs are reported for members of the Safety Population: all participants who applied ruxolitinib cream or vehicle cream at least once. For the Treatment-Extension (TE) Period, TEAEs are reported for the TE Evaluable Population: all participants who applied ruxolitinib cream at least once in the TE Period.
Groups:
- Vehicle Cream BID: Participants applied matching vehicle cream twice a day (BID) for 24 weeks in the Double-Blind Period.
- Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib cream during the Double-Blind Treatment Period and the Treatment-Extension Period. Participants applied ruxolitinib 1.5% cream BID for 24 weeks. Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-Blind Period continued to apply ruxolitinib cream 1.5% BID for an additional 28 weeks in the Treatment-Extension Period. Participants who applied vehicle cream BID during the Double-Blind Period applied ruxolitinib cream 1.5% BID for 28 weeks in the Treatment-Extension Period.
Arm/Group | Vehicle Cream BID | Ruxolitinib Cream 1.5% BID
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/326
Serious Adverse Events (participants affected / at risk) | 0/115 | 6/326
Other Adverse Events (participants affected / at risk) | 6/115 | 56/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=115) | Ruxolitinib Cream 1.5% BID (N=326)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=115) | Ruxolitinib Cream 1.5% BID (N=326)
Application site acne (General disorders) | 3 (3) | 20 (24)
COVID-19 (Infections and infestations) | 2 (2) | 24 (25)
Nasopharyngitis (Infections and infestations) | 1 (1) | 17 (17)

LIMITATIONS AND CAVEATS:
Data from participants at a single site were excluded from all efficacy analyses done on the Intent-to-Treat Population owing to serious noncompliance with the protocol resulting in serious concerns with the data quality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2019-06-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04057573/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04057573/SAP_001.pdf